CLINICAL TRIAL: NCT02798783
Title: Enlarged Vestibular Aqueduct Patient Registry at University Hospitals Rainbow Babies and Children's Hospital
Brief Title: Enlarged Vestibular Aqueduct Registry
Acronym: EVAR
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-16-06
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Enlarged Vestibular Aqueduct; Sensorineural Hearing Loss
Keywords: Vestibular Aqueduct; SLC26A4; FOXI1; Temporal Bone
MeSH Terms: conditions — Deafness, Autosomal Recessive 4; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnosed with EVA: Self-reported Enlarged Vestibular Aqueduct (EVA), or, when available, radiological diagnosis of EVA will be used to define the cohort.

SUMMARY:
People with the congenital anatomical malformation known as "Enlarged Vestibular Aqueduct" (EVA) may experience decline in hearing ability. This is an online registry to gather patient experiences with EVA, with the goal of providing future researchers with the information necessary to better evaluate and make recommendations for patients with EVA. Data will be obtained from volunteers who enroll and submit their information on a website, https://eva.uhhospitals.org, and a limited data set may be provided to researchers interested in analyzing repository data. The limited data set would not contain any identifiable information except for ages, dates such as date of diagnosis, or city/state of residence.

EVA Research Project Website: http://rainbow.org/EVAResearch

EVA Patient Registry Website: https://eva.uhhospitals.org

DETAILED DESCRIPTION:
Study design

The present study would employ a prospective questionnaire and retrospective chart review to develop a centralized registry of EVA patient information. The questionnaire would be administered using custom-designed software and an internet web site that uses secure information transfer protocol and encryption. Given authorization for the release of Protected Health Information (PHI), respective clinicians would be contacted for medical records that would be entered alongside corresponding self-reported data. Interested researchers will be allowed to obtain data, given their respective institution's Institutional Review Board (IRB) approval and documentation thereof. The study would initially continue for four years, and continue based on enrollment numbers and data requests.

Study procedure

Collection methods would be chosen by the participant, and can include one or both of a questionnaire and/or Authorization for the Release of PHI and relevant medical records retrieval.

Implementation of this project would involve three separate components: participant data collection and interaction, (if authorized) PHI retrieval, and data provision to interested researchers.

Questionnaire Data Collection

Upon providing an electronic signature, participants will be taken to a page where they can begin the questionnaire. Patients who begin the questionnaire will be presented with web pages asking for history relating to EVA. Please note that these web pages all offer the option to exit the questionnaire. Patients who elect to provide the Authorization for the Release of PHI will be provided the form to print and mail to the study center (University Hospitals Case Medical Center).

Clinical Data Retrieval and Data Quality

For those participants who do provide Authorization for the Release of PHI, the clinicians whose information was included on the authorization form will be contacted and information requested. This process would involve a transfer of the Authorization for the Release of PHI in one of two ways: either by mail, or via fax. Clinicians who are willing to provide information will be instructed to transmit, via fax or mail, health data to the otolaryngology department at University Hospitals.

Health data that is received will be reviewed and input into forms similar to those that the patients fill. Such a mechanism will provide redundancy to data provided by participants, thus ensuring the quality of this data.

Providing Data to Researchers

The data that is collected will cover a range of topics related to EVA, and will be held with the aim of providing subsets of the data to interested researchers who have IRB approval from their own institutions. A form on the website will list fields for interested researchers to complete, including upload of an IRB protocol. Interested researchers would also be required to complete a Data Use Agreement.

Informed consent procedure

Consent will be obtained electronically and stored separately from patient data, such that identifiable information will only be linked to healthcare data using a patient identification (ID) number.

Potential participants who elect to visit the EVAR website would be presented with an option to participate in the EVAR. From there, participants would be directed to an informed consent web page that contains all of the same information that would be in a written informed consent, a blank version of which is provided in attached documents. The web site would have a field where participants can type their name and the date to signify consent, and another field where participants (if applicable) can type their name and the date to signify assent. Completion of such a field would be considered equivalent to written consent, and is referred to in this document as an "electronic signature".

Only after completing an electronic consent would potential participants be allowed to share questionnaire or authorization information. This means that before seeing the questionnaire or authorization for the release of protected health information, the participant would be required to provide electronic consent.

The consent document itself would be provided to all potential participants, in the form of a downloadable Portable Document Format (PDF) file and as a separate html web page that does not have a section where consent may be entered. This twofold approach will ensure that potential participants can both view the consent in their web browser using the html version, and print the PDF consent in the format that it was accepted by the University Hospitals IRB.

Authorization to Release PHI Procedure

After providing an electronic signature for the informed consent, participants will have the opportunity to complete an Authorization to Release PHI form. Please see attachments for an example of this form.

Participants who provide the information necessary to fill this form would be given the option of printing the form for themselves, or receiving the form in the mail with return postage. In either case, the form would be populated with participant-provided data and provided such that only a participant signature and date would be needed to complete the form. For participants who elect to receive the form in the mail, two copies would be provided to allow the participant to keep one. In either case, participants would be asked to sign and date the document and mail it to the Otolaryngology Department at University Hospitals Case Medical Center (UHCMC). Original documents would be copied and, along with the copy, stored in a locked cabinet that is in a normally locked office on the UHCMC campus.

Data security

Data transfer will occur using secure internet protocol, using computers physically located on a University Hospitals campus.Participant information will be maintained in a secure, HIPAA-compliant server located on a University Hospitals campus. Only database developers and study personnel will have access to this data. For patients who provide Authorization to release PHI, data will only be received via fax, mail, or through University Hospitals email, and will be stored on secure University Hospitals servers.

Identifiable information will be protected from improper use or disclosure by storing data on a secure server located on the University Hospitals campus. When submitting data over the internet, participants will be connecting directly with University Hospitals servers using secure https protocol such that there will be no data access to anyone outside of the participant and server.

For patients who provide Authorization to release PHI, data will only be received via fax, mail, or through University Hospitals email.

Identifiable information will not be reused or disclosed to any other person or entity outside University Hospitals other than those identified in the protocol, except as required by law, for authorized oversight of this research study, or as specifically approved for use in another study by an IRB. Any access to the website or data itself will be reviewed on a monthly basis.

Statistical analysis and sample size calculations

Data on such a wide variety of patient experience measures is unavailable to determine effect sizes and subsequent minimum sample sizes, particularly for an end-point with likely high variability such as self-reported hearing loss. For this reason, and to ensure greatest possible discrimination of effects, the EVA registry will be open to as many people as are willing to enroll. Previously, a mailing list for interested participants was created, and 53 people signed up over the course of three weeks. Sizes of online special interest groups (such as the Yahoo group, http://health.groups.yahoo.com/group/LVAS) have between 1000 and 3000 registered users. Given mailing list interest, and other online community sizes, the investigators expect 300 participants to enroll.

Statistical methods will be left to researchers who request this data, but the data has been organized to facilitate descriptive and model-based statistical characterization of the EVA population. Hearing loss progression may be evaluated in multiple dimensions, particularly in relation to events such as head trauma or flying. For example, such categories of treatment (head trauma, flying) are amenable to analysis with respect to outcomes (hearing loss progression) by such tests as the Chi-square test. Other researchers may be interested in understanding the time taken to diagnose EVA, in which case the interval between date of birth and date of first imaging study can be modeled with respect to other available data points.

Data elements to be collected:

Part 1 - Demographics:

* Relationship of respondent to patient
* Patient:
* Date of Birth
* Gender
* City
* State
* Guardian:
* Date of Birth
* Gender
* City
* State
* Contact:
* Email
* Phone

Part 2 - Initial Findings

* Age at diagnosis of hearing loss
* Diagnostic method
* Audiogram, Otoacoustic Emissions Testing, Auditory Brainstem Response, or other?
* Age at first imaging study
* First image type
* Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)?
* Imaging results
* Which ear has EVA
* Left, right, or both
* Diameter of the vestibular aqueduct

Part 3 - Progression

* Has there been progression of hearing loss?
* Date and age of progression of hearing loss diagnosis - also, commands?
* Events that contributed to hearing loss, open text box
* Did the family notice hearing loss or its event
* Was the hearing loss recognized coincidentally on a hearing screen/routine audiogram?
* Was the patient treated for hearing loss?
* Check boxes for treatment with steroids or other

Part 4 - Trauma and Flying

* Has the patient had any documented head trauma?
* Date and age of trauma - also, commands?
* Was there any associated hearing loss?
* What additional testing was performed, if any?
* Was additional imaging done?
* Has the patient flown?
* Was there any subjective worsening of hearing?
* Was additional testing required after flying?

Part 5 - Family History

* Is there any family history of hearing loss?
* Is there any family history of EVA?
* Has any genetics testing been completed?
* If so, what type of testing?
* At what age?
* What were the results?
* Does the patient have Pendred syndrome?

Part 6 - Aids

* Does the patient receive speech therapy?
* If so, how often?
* At what age did speech therapy begin?
* Does the patient use a Frequency Modulation (FM) system at school?
* Does the patient use a hearing aid?
* If so, in which ear?
* Starting at what year of age?
* Does the patient have a cochlear implant?
* If so, in which ear?
* What year was the operation performed?
* If two implants, were they done at the same time?
* At what age was the operation performed?
* How long after diagnosis of hearing loss was the operation performed?
* How long after diagnosis of EVA was the operation performed?

Part 7 - Vertigo

* Has the patient ever had balance problems or vertigo?
* If so, how frequently?
* How severe?
* Are there triggering activities?
* At what age was the first episode?
* How long after diagnosis did vertigo occur?

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of Enlarged Vestibular Aqueduct OR
* Radiological diagnosis of Enlarged Vestibular Aqueduct

Exclusion criteria:

* None

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes those people who report having a diagnosis of Enlarged Vestibular Aqueduct. The cohort will be defined by voluntary submission of information to a website, eva.uhhospitals.org.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Self-reported lifelong hearing loss progression, subjectively as a questionnaire response and as hearing thresholds (dB) change in clinical documentation. | Through study completion, an average of one year
  Patients will be asked about the progression of hearing loss, including the date and age at which hearing loss progressed. This will be clinically corroborated by evaluating hearing threshold changes via clinical documentation (e.g. audiogram, OAE, ABR)

SECONDARY OUTCOMES:
Age in years at diagnosis of hearing loss, subjectively as a questionnaire response and in clinical documentation. | Through study completion, an average of one year
  Participants will be asked about age at which hearing loss occurred and corroborated by clinical documentation of hearing loss.
Age in years at first CT or MRI used to diagnose Enlarged Vestibular Aqueduct, subjectively as a questionnaire response and in clinical documentation. | Through study completion, an average of one year
  Patients will be asked to specify the age and type of imaging used to diagnose EVA. Participant medical charts and clinical documents (e.g. radiological imaging impressions) will be used to evaluate the presence of EVA and diameter of the vestibular aqueduct in each affected ear.
Hearing loss progression after flying on an airplane, subjectively as a questionnaire response and as hearing thresholds (dB) change in clinical documentation | Within four weeks of flight travel
  Patients will be asked about hearing loss progression after flying on an airplane. If additional testing was done to confirm hearing loss progression, this will be recorded.
Use of hearing aids, subjectively as a questionnaire response or as recorded in prior clinical documentation. | Through study completion, an average of one year
  Participants will be asked about hearing therapies, including use of hearing aids, speech therapy, FM systems in school, and cochlear implantation. If provided, participant medical charts will also be reviewed to determine use of hearing aids.
Hearing loss progression after documented head trauma, subjectively as a questionnaire response or as recorded in prior clinical documentation. | Within four weeks of head trauma
  Participants will be asked about hearing loss progression following a documented head trauma, including the date and age of trauma. If additional testing was done to confirm hearing loss progression, this will be recorded.
Family history of hearing loss, subjectively as a questionnaire response or as recorded in prior clinical documentation. | Through study completion, an average of one year
  Patients will be asked about family history of hearing loss, including any genetic testing that has been completed.
Balance problems or vertigo, subjectively as a questionnaire response or as recorded in prior clinical documentation. | Through study completion, an average of one year
  Patients will be asked about problems they've experienced related to vertigo and balance problems, including the frequency, severity, activities that may have triggered it, age of first episode, and how long vertigo occurred after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Otteson, MD, MPH, Principal Investigator — University Hospitals Cleveland Medical Center; Cliff Megerian, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Benjamin A Reinthal, Study Director — University Hospitals Cleveland Medical Center; Mustafa S Ascha, MS, Study Director — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited data set will be available to researchers who demonstrate IRB approval for a study that would require the use of data points collected by the Enlarged Vestibular Aqueduct Registry. This dataset will include information only in accordance with HIPAA definitions of a limited dataset, for example, excluding names and addresses. Data will be available one year after enrollment is to start, on June 2, 2017. The data may be obtained by submission of a request along with proof of investigator institutional review board approval, forms for which will be available through the registry web site.
Time Frame: Data will be available one year after enrollment is to start, on June 2, 2017. The study would initially continue for four years, and continue based on enrollment numbers and data requests.
Access Criteria: Background information:
  * Corresponding researcher
  * Name
  * Title
  * Institution
  * Department
  * Address
  * Contact phone number
  * Contact email address
  * Principal Investigator
  * Name
  * Title
  * Institution
  * Department
  * Address
  * Contact phone number
  * Contact email address
  * Origin of the protocol (e.g. investigator-initiated, industry, federal agency, cooperative group, other)
  Study information:
  * Full title of study
  * Whether the research has IRB approval
  * Background/rationale/significance
  * Purpose/Hypothesis
  Document Upload:
  * Approved IRB Protocol Application
  * Signed CV for each investigator listed on the IRB application
  * Signed Data Use Agreement

REFERENCES:
- [Background] Valvassori GE, Clemis JD. The large vestibular aqueduct syndrome. Laryngoscope. 1978 May;88(5):723-8. doi: 10.1002/lary.1978.88.5.723. PMID 306012
- [Background] Gopen Q, Zhou G, Whittemore K, Kenna M. Enlarged vestibular aqueduct: review of controversial aspects. Laryngoscope. 2011 Sep;121(9):1971-8. doi: 10.1002/lary.22083. Epub 2011 Aug 16. PMID 22024854
- [Background] Griffith AJ, Wangemann P. Hearing loss associated with enlargement of the vestibular aqueduct: mechanistic insights from clinical phenotypes, genotypes, and mouse models. Hear Res. 2011 Nov;281(1-2):11-7. doi: 10.1016/j.heares.2011.05.009. Epub 2011 Jun 6. PMID 21669267
- [Background] Madden C, Halsted M, Benton C, Greinwald J, Choo D. Enlarged vestibular aqueduct syndrome in the pediatric population. Otol Neurotol. 2003 Jul;24(4):625-32. doi: 10.1097/00129492-200307000-00016. PMID 12851556
- [Background] Dewan K, Wippold FJ 2nd, Lieu JE. Enlarged vestibular aqueduct in pediatric sensorineural hearing loss. Otolaryngol Head Neck Surg. 2009 Apr;140(4):552-8. doi: 10.1016/j.otohns.2008.12.035. PMID 19328346
- See also: The EVA Patient Registry Website — https://eva.uhhospitals.org
- See also: The EVA Research Project Website — http://rainbow.org/EVAResearch